CLINICAL TRIAL: NCT03245047
Title: A Prospective Randomized Double Blind Clinical Study to Determine the Clinical Impact of ONS in Community-dwelling Elderly
Brief Title: The Nutritional Health for the Elderly Reference Centre Study (The NHERC Study)
Acronym: NHERC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Collaborators: Changi General Hospital (Other); SingHealth Polyclinics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BL35 (Part 2)
Record Dates: First submitted 2017-08-01; First posted 2017-08-10 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, placebo controlled, double-blind, parallel design, multi-center study. Eligible participants will be randomly allocated to one of two groups: oral nutritional supplement with dietary counseling group or placebo supplement with dietary counseling group. Randomization will be stratified by MUST malnutrition status (medium risk or high risk) and site of recruitment. All participants, including both recently discharged patients from the hospital or elderly recruited from the polyclinics.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is double-blinded, i.e., during the study, neither the investigator(s), study and appropriate Abbott Nutrition staff, nor participants will be informed of the identity of any of the study products. Study center personnel will not analyze the contents of the study products or in any way seek to learn the identity of the study products. The investigator should ensure that if it becomes necessary, blinding is broken only in accordance with the protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Dietary Supplement: Oral Nutritional Supplement with AN777 Participants in the intervention group will be asked to consume two servings of oral nutritional supplement per day for 180 days. (Oral Consumption)
  Interventions: Dietary Supplement: Oral Nutritional Supplement with AN 777
- Control group (Placebo Comparator): Participants in the control group will be asked to consume two servings of Oral nutritional supplement per day for 180 days.(Oral Consumption)
  Interventions: Other: Oral Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: Oral Nutritional Supplement with AN 777 — Oral Nutritional Supplement with AN 777, 2 servings a day
  Arms: Intervention group
Other: Oral Nutritional Supplement — Oral Nutritional Supplement, 2 servings a day
  Arms: Control group

SUMMARY:
The prevalence of malnutrition among the elderly in Asia is high. The objective of this randomized, parallel, placebo controlled, double-blind study is to evaluate the effects of consuming an adult ONS plus dietary counseling (intervention group) for 180 days on nutritional status and unexpected hospital (re)admission, compared with a placebo supplement plus dietary counseling (control group).

DETAILED DESCRIPTION:
This randomized controlled trial will involve 800 elderly who are at risk of undernutrition (MUST score ≥ 1). Participants will be screened for eligibility. Recruitment will be at the polyclinic and in the inpatient ward prior to their discharge from the hospital. Participants will be randomized to intervention group vs. control group at the baseline visit at the clinical trial research unit where baseline measurements and baseline survey using the study specific questionnaires will be performed. Participants will be followed up prospectively at Day 30, Day 90, Day 180 (exit visit), and Day 360 (post-intervention follow-up visit). Repeated measures will be performed at the pre-defined time points. Intention-to-treat analysis comparing intervention group vs. control group will be performed to study the effect of ONS on primary composite outcome consisting of (i) change in body weight from baseline to Day 180 or (ii) unexpected admission to the hospital over 180-day intervention period. The effect of ONS on nutritional status will be examined by comparing the biochemical and anthropometric measurements of intervention group vs. control group at Day 180. Other outcomes such as changes in functional assessment, nutritional knowledge levels, and quality of life will also be examined. There will be a follow up visit at Day 360.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant aged ≥65 years.
2. Community-dweller, i.e. not staying in a residential intermediate and long-term care (ILTC) service institution.
3. Participant is being discharged home directly (applicable for hospital cohort).
4. Participant is community ambulant with or without aid.
5. Participant does not have any chronic disease(s) or has stable chronic disease(s) including hypertension, chronic obstructive pulmonary disease, and cardiovascular disease in the opinion of the Study Physician, at study entry
6. Participant has voluntarily signed and dated an informed consent form (ICF), approved by an Institutional Review Board (IRB) and provided authorization prior to any participation in the study.
7. Participants will be able to communicate and follow instructions.
8. Participant is able to consume food and beverages orally.
9. Participant has been identified as at risk of undernutrition as defined by Malnutrition Universal Screening Tool.
10. Participant is willing to refrain from taking non-study oral nutritional supplements including protein powder over the entire course of the study.
11. Participant is able and willing to follow study procedures and record data in diary and complete any forms or assessments needed throughout the study, with or without the help of the caregivers.

Exclusion Criteria:

1. Participant has been diagnosed with dementia according to medical records.
2. Participant has been diagnosed with type 1 or type 2 diabetes according to medical records. (Note: This includes participant with controlled diabetes.)
3. Participant has any active infectious disease (such as tuberculosis, Hepatitis B or C, HIV infection) according to medical records.
4. Participant has been diagnosed with severe gastrointestinal disorders including celiac disease, short bowel syndrome, pancreatic insufficiency, or cystic fibrosis according to medical records.
5. Participant has been diagnosed with end stage organ or pre-terminal diseases or acute myocardial infarction within the last 30 days from the screening according to medical records.
6. Participant has malignancy according to medical records.
7. Participant has any other clinically significant medical condition, which in the investigator's opinion, makes him or her unsuitable for inclusion in the study.
8. Participant is taking part in another study that has not been approved as a concomitant study by the study team.
9. Participant has been diagnosed or is known to be allergic or intolerant to milk products.
10. Participant has continuous ONS usage for 30 days prior to the screening.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 811 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Primary composite outcome consisting of change in body weight and unexpected hospital admission | baseline to Day 180
  (i) change in body weight from baseline to Day 180 or (ii) unexpected admission to the hospital over 180-day intervention period (Death before any unexpected admission to the hospital will be counted as a hospitalization event)

SECONDARY OUTCOMES:
Fat mass and fat free mass | Baseline, 30 days, 90 days and 180 days]
  Fat mass and fat free mass in kilograms will be measured using Tanita MC-780
Length of stay of unexpected hospital admission(s) | 90 days & 180 days
  Unexpected admission to the hospital over 90-day and 180-day intervention periods

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Siew Ling Tey, Ph.D., Study Chair — Abbott Nutrition Research & Development; Samuel TH Chew, MB.BCh.BAO, Principal Investigator — Changi General Hospital
Locations (4):
- Singapore (4):
  - Marine Parade Polyclinic, Singapore
  - Bedok Polyclinic, Singapore
  - Tampines Polyclinic, Singapore
  - Changi General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chew STH, Tey SL, Yalawar M, Liu Z, Baggs G, How CH, Cheong M, Chow WL, Low YL, Huynh DTT, Tan NC. Prevalence and associated factors of sarcopenia in community-dwelling older adults at risk of malnutrition. BMC Geriatr. 2022 Dec 24;22(1):997. doi: 10.1186/s12877-022-03704-1. PMID 36564733
- [Derived] Chew STH, Tan NC, Cheong M, Oliver J, Baggs G, Choe Y, How CH, Chow WL, Tan CYL, Kwan SC, Husain FS, Low YL, Huynh DTT, Tey SL. Impact of specialized oral nutritional supplement on clinical, nutritional, and functional outcomes: A randomized, placebo-controlled trial in community-dwelling older adults at risk of malnutrition. Clin Nutr. 2021 Apr;40(4):1879-1892. doi: 10.1016/j.clnu.2020.10.015. Epub 2020 Oct 15. PMID 33268143